CLINICAL TRIAL: NCT06571656
Title: Evaluation of the Safety and Tolerability of Ocular Lubricants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DEE253-E002
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye Disease
Keywords: Scratchy eyes; Dry eyes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Other): FID123359/ FID123360/ FID123361/FID121843: One drop in each eye, test formulation or ocular lubricant as randomized, at respective Investigational Product visit. A total of 4 drops per eye will be instilled.
  Interventions: Other: FID123359 test formulation; Other: FID123360 test formulation; Other: FID123361 test formulation; Other: FID121843 ocular lubricant
- Sequence 2 (Other): FID123360/ FID123361/FID121843/ FID123359: One drop in each eye, test formulation or ocular lubricant as randomized, at respective Investigational Product visit. A total of 4 drops per eye will be instilled.
  Interventions: Other: FID123359 test formulation; Other: FID123360 test formulation; Other: FID123361 test formulation; Other: FID121843 ocular lubricant
- Sequence 3 (Other): FID123361/FID121843/FID123359/ FID123360: One drop in each eye, test formulation or ocular lubricant as randomized, at respective Investigational Product visit. A total of 4 drops per eye will be instilled.
  Interventions: Other: FID123359 test formulation; Other: FID123360 test formulation; Other: FID123361 test formulation; Other: FID121843 ocular lubricant
- Sequence 4 (Other): FID121843/FID123359/ FID123360/ FID123361: One drop in each eye, test formulation or ocular lubricant as randomized, at respective Investigational Product visit. A total of 4 drops per eye will be instilled.
  Interventions: Other: FID123359 test formulation; Other: FID123360 test formulation; Other: FID123361 test formulation; Other: FID121843 ocular lubricant

INTERVENTIONS:
Other: FID123359 test formulation — Investigational product
Other: FID123360 test formulation — Investigational product
Other: FID123361 test formulation — Investigational product
Other: FID121843 ocular lubricant — Commercially available, preservative-free eye drops
  Other Names: SYSTANE HYDRATION

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of three new artificial tear formulations in subjects with moderate dry eye disease.

DETAILED DESCRIPTION:
This study will be conducted in 2 stages. In Stage 1, subjects will attend a total of 10 scheduled visits: one Screening visit, four Investigational Product visits, four 12-hour Follow Up visits (one for each Investigational Product visit), and an Exit visit. At each Investigational Product visit, subjects will receive one drop of the investigational product in each eye (2 drops total), as randomized. The first Investigational Product visit will occur 1 to 7 days after the Screening visit. A washout period of 2 to 7 days will separate each Investigational Product visit. Total individual duration of participation in Stage 1 will be 8 to 34 days. The planned enrollment for Stage 1 is 72 subjects.

At the conclusion of Stage 1, an interim analysis will be conducted to help determine potential adaptations to the study design for Stage 2.

This study will be conducted in Australia.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to understand and sign an Ethics Committee-approved informed consent form.
* Willing and able to attend all study visits as required by the protocol.
* Exhibits symptoms of dry eye at the Screening Visit.
* Currently uses habitual artificial tears to alleviate dry eye symptoms.
* Willing and able to maintain similar environmental conditions throughout the study (for example, avoid extreme changes in humidity/temperature, avoid windy conditions) and refrain from swimming on Investigational Product visit days.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Has any known active ocular disease and/or infection.
* Has any known infection or inflammation that requires treatment or has a systemic condition that in the opinion of the investigator, may affect a study outcome variable.
* Has had an ocular injury to either eye in the past 12 weeks prior to screening.
* Currently wears contact lenses or has a history of contact lens wear within the previous 1 month.
* Has undergone any ocular surgery (including intraocular surgery) within the past 12 months or has any ocular surgery planned during the study.
* Is pregnant, intends to become pregnant, or is breastfeeding.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (AEs) | Visit 2 (1 to 7 days after the Screening Visit) through Visit 6/Study Exit. Visit 6 will occur 7 to 27 days after Visit 2 depending on observed visit windows.
  An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). The number of adverse events as observed or reported will be recorded.
Number of Subjects with Biomicroscopy Findings Outside of Normal Limit | Screening Visit through Visit 6/Study Exit. Visit 6 will occur 8 to 34 days after Screening Visit, based on observed visit windows.
  The investigator will observe the corneal and other ocular structures under white light of the slit lamp. The number of subjects with biomicroscopy findings outside of normal limits will be recorded.
Best Corrected Visual Acuity (BCVA) | Screening through Visit 6/Study Exit. Visit 6 will occur 8 to 34 days after Screening Visit, based on observed visit windows.
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) letter charts and recorded in logarithm Minimum angle of resolution (logMar).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Dry Eye, Study Director — Alcon Research, LLC
Locations (5):
- Australia (5):
  - School of Optometry and Vision, Sydney, New South Wales
  - Advanced Optometry, Spring Hill, Queensland
  - Ophthalmic Trials Australia, Teneriffe, Queensland
  - The University of Melbourne, Department of Optometry and Vision Science, Carlton, Victoria
  - Deakin Collaborative Eye Care Clinic, Waurn Ponds, Victoria

IPD SHARING:
Plan to Share IPD: No